CLINICAL TRIAL: NCT07146893
Title: Feasibility Study for Repurposing RET Inhibitors for Treating Cancer Cachexia
Brief Title: Feasibility Study for Repurposing RET Inhibitors
Acronym: FEATHER
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Presbyterian Health Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-FEATHER; PHF-CTGA (Other: Presbyterian Health Foundation)
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cachexia-Anorexia Syndrome
Keywords: RET inhibitor
MeSH Terms: interventions — selpercatinib

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm feasibility study to assess the effects of selpercatinib on cachexia and anorexia in patients with NSCLC, colorectal cancer, or pancreatic cancer who are undergoing platinum-based chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Significant Weight Loss (Experimental): Patients will be weighed at baseline, 4, 8, and 12 weeks while on treatment and again at the 16-weeks after treatment has been discontinued to asses for changes in weight.
  Interventions: Drug: Selpercatinib; Other: Strength Assessment

INTERVENTIONS:
Drug: Selpercatinib — Patients will be instructed to take selpercatinib orally (PO) twice daily (BID), approximately every 12 hours. While on study, they will undergo weight measurements and regular blood draws every 4 weeks. At the 16-week post-treatment follow-up, patients will return to the clinic for a weight assessment to evaluate potential changes in body weight.
  Patients will be administered assessments including, Functional Assessment of Anorexia Cachexia Therapy (FAACT), administered at screening, at 12 weeks post-discontinuation of the study drug, and again at the 16-week follow-up.
  Other Names: RETEVMO
Other: Strength Assessment — Several strength assessment will be conducted at baseline and at 12 weeks end-of-treatment, which will include measurements such as grip strength, hallux strength, timed chair stands, leg press, and localized ultrasound of the quadriceps.

SUMMARY:
The purpose of this study is to assess the effects of selpercatinib on cachexia and anorexia in patients diagnosed with NSCLC, colorectal cancer, or pancreatic cancer.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the feasibility of selpercatinib in addressing cachexia and anorexia among patients with non-small cell lung cancer (NSCLC), colorectal cancer, or pancreatic cancer who are eligible for platinum-based chemotherapy per standard of care. Participants will undergo blood draws at baseline and at 4, 8, and 12 weeks while on selpercatinib. At 16 weeks patients will return to the clinic for a weight assessment.

Study evaluations will include the Functional Assessment of Anorexia Cachexia Therapy (FAACT), administered at screening, at 12 weeks post-discontinuation of the study drug, and again at the 16-week follow-up. In addition, several assessments of overall muscle strength and function will be conducted including a hallux strength assessment, sub-maximal leg press, sit-to-stand timing, grip strength, and ultrasound of the quadriceps. These will be conducted at baseline and again at 12 weeks end-of-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and documented locally advanced or metastatic NSCLC, pancreatic ductal adenocarcinoma, or colorectal cancer
* Patient is currently receiving platinum-based therapy for cancer treatment
* Patients on stable EPI
* Written informed consent signed and dated by the patient prior to the performance of any study-specific procedures, sampling, or analyses
* At least 18 years-of-age at the time of signature of the informed consent form (ICF)
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2
* Plasma GDF-15 level is at least 1500pg/mL
* Life expectancy exceeds 4 months, as judged by investigator
* Cachexia, defined as weight loss of >5% body weight in the past 6 months, OR weight loss of >2% body weight in the past 6 months with BMI < 20

Exclusion Criteria:

* ECOG Performance Score of 3 or 4
* Is pregnant or plans to become pregnant during study duration (if patient is of childbearing potential) or plans to make someone pregnant during study duration.
* Patient has not experienced significant weight loss (defined as loss of >5% body weight in the past 6 months, OR loss of >2% body weight in the past 6 months with BMI < 20)†
* Out-of-range laboratory values defined as:

  * Absolute neutrophil count (ANC) <1.5 x 109/L
  * Hemoglobin (Hgb)90 g/L or <9 g/dL
  * Platelets <100 x 109/L
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2.5 x the upper limit of normal (ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
  * Total bilirubin >1.5 x ULN (unless the patient has Grade 1 bilirubin elevation due to Gilbert's disease or a similar syndrome involving slow conjugation of bilirubin)
  * Creatinine >1.5 times ULN (patients may enter if creatinine is >1.5 x ULN and estimated glomerular filtration rate (eGFR) is >30 mL/min/1.73 m2 according to the Chronic Kidney Disease Epidemiology Collaboration equation); confirmation of eGFR is only required when creatinine is >1.5 X ULN
  * International Normalization Ratio (INR) >2
* Ongoing treatment with anti-seizure medications that induce the CYP3A enzyme
* Presence of active gastrointestinal disease or other conditions that will interfere significantly with the absorption, distribution, metabolism, or excretion of selpercatinib(e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea Grade ≥2)
* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, uncontrolled diabetes mellitus, active bleeding diatheses, or active infection including hepatitis B, hepatitis C, and human immunodeficiency virus. Screening for chronic conditions is not required.
* Presence of other active invasive cancers other than the ones treated in this study within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin, or in situ carcinoma of uterine cervix, or other local tumors considered cured by local treatment.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol.
* Pneumonitis or QTc prolongation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2026-02-26 (Estimated); Primary Completion 2027-02-23 (Estimated); Study Completion 2028-02-23 (Estimated)

PRIMARY OUTCOMES:
Mean (± SD) changes in body weight after 12 weeks | 12 weeks
  At screening, patients will have their initial weight recorded. While on study, they will take selpercatinib orally twice daily, with weight assessments conducted every four weeks (Weeks 4, 8, and 12). Selpercatinib will be discontinued at Week 12, and at the 16-week post-treatment follow-up, patients will return to the clinic for a final weight assessment.
Mean (± SD) percentage of doses of selpercatinib taken on time by patient | 12 weeks
  A pill diary will be provided to patients to record the time, date, and dose (40 mg or 80 mg) of selpercatinib before starting the study drug.

SECONDARY OUTCOMES:
Mean (± SD) changes in anorexic behaviors after 12 weeks | 12 weeks
  Patients will be administered a Functional Assessment of Anorexia Cachexia- Anorexia Cachexia Subscale (FAACT-ACS) at baseline, and again at 12 weeks. The FAACT-ACS is designed to assess patient well-being and concerns using a Likert scale, where responses range from 0 to 4. A score of 0 indicates "Not at all," representing the lowest level of agreement or concern, while a score of 4 indicates "Very much," representing the highest level.
Mean (± SD) changes in skeletal muscle while taking selpercatinib | 12 Weeks
  Regular blood draws every 4 weeks while on selpercatinib will be taken with the goal of quantifying GDF-15 levels in each patient. Also a lumbar muscle assessment using a CT scan at baseline and again at 12 weeks to assess for muscle changes while taking selpercatinib.
Mean (± SD) changes in Strength outcomes in patients taking selpercatinib | 12 weeks
  A Hallux Strength Test will be conducted at baseline and repeated at 12 weeks (+/- 2 weeks), measuring grip strength, timed chair stands, leg press, and localized ultrasound of the quadriceps.
Mean (± SD) changes in plasma GDF-15 while taking selpercatinib | 12 Weeks
  Regular blood draws every 4 weeks while on selpercatinib will be taken with the goal of quantifying GDF-15 levels in each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Nirmal Choradia, MD, Principal Investigator — University of Oklahoma - Stephenson Cancer Center
Locations (1):
- OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No